CLINICAL TRIAL: NCT00975494
Title: Chronic PDE5-Inhibition With Sildenafil Improves Diastolic Function, Cardiac Geometry and Clinical Status in Patients With Stable HF: A 1-Year Prospective Randomized, Placebo-Controlled Study
Brief Title: Chronic Sildenafil Treatment in Heart Failure
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Milan (Other)
Responsible Party: Marco Guazzi (PI), University of Milano, Cardiology
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 444-05
Record Dates: First submitted 2009-09-03; First posted 2009-09-11 (Estimated); Last update posted 2009-09-11 (Estimated); Status verified 2009-09

CONDITIONS: Heart Failure
Keywords: pde5-inhibition; sildenafil; LV diastolic function; heart failure patients
MeSH Terms: conditions — Heart Failure | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- sildenafil (Active Comparator): sildenafil 50 mg three times/day
  Interventions: Drug: Sildenafil
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sildenafil
  Arms: sildenafil
Drug: Placebo
  Arms: Placebo

SUMMARY:
In heart failure (HF), a defective nitric oxide (NO) signaling may be involved in left ventricular (LV) diastolic abnormalities and LV remodelling progression. PDE5-inhibition, by blocking NO degradation and overexpressing cellular cyclic guanosine monophosphate (cGMP) pathways might be beneficial. Several short term studies have demonstrated safety and clinical improvement in stable heart failure (HF) patients.

The purpose of this study is to test the effects on LV diastolic function, cardiac geometry and clinical status in a cohort of HF patients.

DETAILED DESCRIPTION:
Heart failure (HF) is a significant health care concern that is evolving to epidemic proportions. Development of new forms of interventions remains a challenging task. An abnormal nitric oxide (NO) pathway is involved in several basic pathophysiological abnormalities encountered in HF syndrome and NO overexpression may represent a desirable therapeutic target in the cure of the disease.

PDE5-inhibition is an intriguing pharmacological strategy to enhance in vivo nitric oxide (NO) signaling by increasing the cyclic guanosine monophosphate (cGMP). availability. A number of theoretical backgrounds support the use of PDE5-inhibitors in HF and an increasing number of clinical studies have been testing PDE5-inhibition as a potential valid adjunct in the management of HF patients.

In failing hearts of animal models, PDE5-inhibition has also provided the attractive therapeutic properties to reverse left ventricular chamber remodelling by preventing and reversing LV cardiac hypertrophy and fibrosis and by protecting the myocardium from ischemia-reperfusion injury and apoptosis. There is also evidence that a defective NO activity plays an important role in the excitation-relaxation process of the failing heart, an effect explained by a defective cGMP-induced phosphorylation of troponin I, which facilitates calcium-independent diastolic cross-bridge cycling and concomitant myocardium diastolic stiffening.

No report has so far investigated whether cardiac function and, primarily, diastolic LV function may be a target of chronic PDE5-inhibition and whether any improvement in diastolic function is related to a reverse effect in cardiac geometry in patients with HF. Furthermore, it is undefined whether a favourable effect on left ventricular function may be involved in the reported changes in important clinical correlates such as functional status and quality of life. We tested these hypotheses, by addressing the effects of chronic sildenafil administration (50 mg three times/day) on diastolic function and clinical status by Tissue Doppler imaging, cardiopulmonary exercise testing and quality of life score.

ELIGIBILITY:
Inclusion Criteria:

* consent to participate in the study after detailed information about procedures, possible clinical benefits and risks;
* negative exercise stress test prior to study initiation;
* forced expiratory volume in 1 sec/forced vital capacity ratio>70%;
* left ventricular ejection fraction < 45%, determined by echocardiography.

Exclusion Criteria:

* subjects unable to complete a maximal exercise test
* systolic blood pressure > 140 and <110 mmHg
* diabetes mellitus
* therapy with nitrate preparations
* history of sildenafil intolerance
* significant lung or valvular diseases
* neuromuscular disorders, claudication
* peripheral vascular disease

Ages: 38 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2005-04; Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Left ventricular diastolic function | 1 year

SECONDARY OUTCOMES:
Functional capacity | 1 year
Quality of life | 1 year
Neurohumoral (brain natriuretic peptide) | 1 year
Cardiac remodeling | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- University of Milano, Milan, Italy

REFERENCES:
- [Derived] Guazzi M, Vicenzi M, Arena R, Guazzi MD. PDE5 inhibition with sildenafil improves left ventricular diastolic function, cardiac geometry, and clinical status in patients with stable systolic heart failure: results of a 1-year, prospective, randomized, placebo-controlled study. Circ Heart Fail. 2011 Jan;4(1):8-17. doi: 10.1161/CIRCHEARTFAILURE.110.944694. Epub 2010 Oct 29. PMID 21036891